CLINICAL TRIAL: NCT05327465
Title: Exercise to Enhance Cardiovascular Health Among Black Prostate Cancer Patients With Androgen Deprivation Therapy: POWER Trial
Brief Title: Exercise to Enhance Cardiovascular Health Among Black Prostate Cancer Patients With Androgen Deprivation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Pfizer (Industry); Prostate Cancer Foundation (Other)
Responsible Party: Principal Investigator, Christina Dieli-Conwright, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-741
Record Dates: First submitted 2022-03-16; First posted 2022-04-14 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Androgen Deprivation Therapy; Prostate Cancer; Prostate Cancer Metastatic
Keywords: Androgen deprivation therapy; Localized Prostate Cancer; Prostate Cancer Metastatic; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic and resistance exercise (Experimental): Virtually supervised 16-week aerobic and resistance exercise performed at home via Zoom.
  The exercises will be performed three times per week for 16 weeks, and virtually supervised by a professional exercise trainer.
  Interventions: Other: Aerobic and resistance exercise
- Usual care (Active Comparator): Maintenance of baseline exercise levels for 16 weeks with an offer to perform the same exercise program after 16 weeks.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Aerobic and resistance exercise — Perform exercise at home with virtual supervision, including aerobic exercise (e.g.,cycling), which can improve cardiovascular (heart) and lung function, and resistance exercise (e.g., dumbbell lifting and using resistance band. The exercises will be performed three times per week for 16 weeks, and virtually supervised by a professional exercise trainer
  Arms: Aerobic and resistance exercise
Other: Usual Care — Maintenance of baseline exercise levels for 16 weeks with an offer to perform the same exercise (aerobic and resistance exercise) program after 16 weeks.
  Arms: Usual care

SUMMARY:
The purpose of this research is to determine whether a 16-week culturally tailored, technology-based, aerobic and resistance exercise intervention improves cardiovascular risk factors in Black men diagnosed with prostate cancer and are undergoing androgen deprivation therapy (ADT), and whether it will also improve physical fitness and function, body composition, and outcomes such as quality of life, cancer symptoms, and self-esteem.

Participants in this study will be randomly assigned to one of two groups: 1) Aerobic and resistance exercise, or 2) Usual care.

DETAILED DESCRIPTION:
The research study procedures include: screening for eligibility, study intervention, and evaluation of blood markers (blood draw), body composition, cardiorespiratory fitness, muscular strength, and surveys at study entry and follow-up visit.

Participants in this study will be randomly assigned to one of two groups: 1) Aerobic and resistance exercise, or 2) Usual care.

* Aerobic and resistance exercise - virtually supervised 16-week aerobic and resistance exercise performed at home via Zoom.The exercise group will be asked to perform exercise at home with virtual supervision, including aerobic exercise. The exercises will be performed three times per week for 16 weeks, and virtually supervised by a professional exercise trainer.
* Usual care - maintenance of baseline exercise levels for 16 weeks with an offer to perform the same exercise program after 16 weeks. The usual care group will be asked to maintain their current exercise levels and will be offered the same exercise intervention after the completion of the study.

All participants will undergo two testing visits throughout the 16-weeks of the study period, with the exercise group part-taking in 1 additional testing visit at week 8 to assess aerobic fitness and muscular strength only.

Participants will be on the research study for 4 months. It is expected that about 62 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all criteria to be eligible, including travel to Dana-Farber Cancer Institute (DFCI) to collect research data to address the study question.
* Over 18 years old; children under the age of 18 will be excluded due to the rarity of the disease
* Histologically diagnosed of localized or metastatic prostate cancer
* Have been receiving androgen deprivation therapy (ADT) (i.e., luteinizing hormone-releasing hormone [LHRH] agonist/antagonist and/or androgen receptor [AR] agonist/antagonist) for at least one month with a plan to continue ADT for at least 4 months at the time of recruitment
* Self-identify as Black
* Medically cleared to participate in exercise by their referred physician or a certified clinical exercise physiologist
* Are without medical conditions that could exacerbate with exercise, such as bone disease (excluding bone metastases) at imminent risk of fracture or uncontrolled cardiopulmonary or metabolic diseases
* Speak English and/or Spanish
* Currently participate in less than or equal to 60 minutes of moderate or vigorous structured exercise/week
* Willing to travel to DFCI for necessary data collection
* Ability to communicate and complete written forms in English and/or Spanish

Exclusion Criteria:

* Are not receiving ADT (i.e., LHRH agonist/antagonist and/or AR agonist/antagonist)
* Pre-existing medical conditions such as uncontrolled cardiopulmonary disease, or metabolic diseases that could exacerbate with exercise
* Are not English or Spanish speaking
* Patients with secondary diagnosis (with the exception of basal cell carcinoma)
* Participate in more than 60 minutes of moderate or vigorous structured exercise/week
* Unable to travel to DFCI for necessary data collection
* May not be able to comply with the safety monitoring requirements of the study in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease risk factors | baseline to 4 months
  Framingham Risk Score, an established comprehensive tool for evaluating the risk of developing cardiovascular disease using blood samples (i.e., low-density lipoprotein-cholesterol [LDL-C] or total cholesterol [TC], high-density lipoprotein-cholesterol [HDL-C]), demographic and medical profiles , and lifestyle behaviors (i.e., age, blood pressure, and diabetic and smoking status). The score ranges from -4 to 36 and the 10-year cardiovascular risk will be calculated accordingly (a higher score indicates a higher risk of cardiovascular disease).

SECONDARY OUTCOMES:
Cardiorespiratory capacity | baseline to 4 months
  Cardiorespiratory fitness will be assessed as VO2peak by a graded maximal cycle exercise stress test. VO2peak is defined as the highest values of oxygen uptake averaged among every 15-second interval during the test. VO2peak will be reported in both relative (ml·kg-1·min-1) and absolute (L/min) terms
Muscular strength | baseline to 4 months
  Muscular strength will be measured as 1-repetition maximum (RM) (i.e., the greatest resistance that can be moved through the full range of motion), which has been the standard for strength assessments. 1-RM values will be estimated from 10-RM using validated equations on 12 exercises including the ten exercises utilized in the prescription not performed on machines.
Short Physical Performance Battery (SPPB) | baseline to 4 months
  Physical function will be assessed by the SPPB. This includes the following 3 lower extremity measures completed in the following order. Timed balance (seconds): Balance will be assessed under 3 conditions (side-by-side, semi-tandem, and tandem stands). Gait speed (seconds): Gait speed will be assessed over a 4-meter flat surface distance. The participant will be asked to complete 2 attempts of this test. Time will be recorded using an electronic timing system. Chair stand (seconds): Chair stand will be performed under 2 conditions: a) subjects will perform a single chair stand; b) subjects will be asked to perform 5 repeated chair stands as quickly as possible; time to completion will be recorded.
Timed-Up-and-Go (TUG) | baseline to 4 months
  Mobility will be assessed using the Timed Up and Go (TUG) test, which has been shown to predict immediate fall risk better than static balance tests or isometric muscle strength. Participants begin seated in a chair with hands on the armrests, are asked to rise, walk to a line on the floor 3 m from the chair, turn around, and return to the same seated position as quickly and safe as possible. Scores will be taken as the time (seconds) to complete the task, with one practice trial given. An average of time for 3 trials is calculated.
Hand grip strength | baseline to 4 months
  Grip strength will be measured using a hand-held dynamometer on the participant's dominant hand. The subject will be asked to grip the handle of the dynamometer with one hand using as much grip pressure (kg) as possible while holding for 2 seconds. The subject will be asked to complete 2 grip strength attempts.
Fat mass | baseline to 4 months
  Fat mass (kg) will be obtained from a whole-body dual-energy x-ray absorptiometry scan (DXA; Lunar DPX-IQ), which provides highly accurate results compared to computed tomography, a gold standard measure of body composition.
Percent body fat | baseline to 4 months
  Percent body fat will be obtained from a whole-body dual-energy x-ray absorptiometry scan (DXA; Lunar DPX-IQ), which provides highly accurate results compared to computed tomography, a gold standard measure of body composition.
Lean mass | baseline to 4 months
  Lean mass (kg) will be obtained from a whole-body dual-energy x-ray absorptiometry scan (DXA; Lunar DPX-IQ), which provides highly accurate results compared to computed tomography, a gold standard measure of body composition.
Hip circumference | baseline to 4 months
  A constant-tension tape measure will be used to obtain waist circumference (i.e., the distance around the waist using the umbilicus as the reference point) (cm).
Waist circumference | baseline to 4 months
  A constant-tension tape measure will be used to obtain hip circumference (the distance around the widest girth of the buttocks using the greater trochanter as a landmark) (cm).
Health-related quality of life - EORTC-QLQ C30 | baseline to 4 months
  European Organization for Research and Treatment of Cancer- Quality of Life Questionnaire-C30 will assess health-related quality of life, consisting of substacles including functional scales (physical, role, cognitive, emotional, social), symptom scales (fatigue, pain, and nausea and vomiting), global health status and quality of life scale, also several single-item symptom measures. The score ranges from 0 to 100 and a higher value indicates a better quality of life.
Prostate cancer-specific symptoms - EPIC-26 | baseline to 4 months
  Expanded Prostate Cancer Index Composite-26 will assess prostate cancer-specific symptoms (e.g., urinary incontinence, sexual dysfunction, and bowel dysfunction). The score ranges from 0 to 100 and a higher value indicates a worse symptom.
Cancer treatment symptoms - MDASI | baseline to 4 months
  MD Anderson Symptom Inventory will assess cancer treatment symptoms (e.g., pain, neuropathy). The score ranges from 0 to 10 and a higher value indicates a worse symptom.
Self-esteem - RSES | baseline to 4 months
  The Rosenberg Self-Esteem Scale will assess self-esteem. The score ranges from 10 to 40 and a higher value indicates a better self-esteem.
Percieved implementation outcomes assessed by AIM, IAM, and FIM | baseline to 4 months
  The Acceptability of Intervention Measure, Intervention Appropriateness Measure, and Feasibility of Intervention Measure will be assessed at post-intervention to measure participant-perceived intervention feasibility and acceptability. Each measure has four items with 5-point likers scale. The values in each measure will be the mean of four items and range from 5-20. A higher value means a more acceptable, appropriate, and feasible intervention, perceived by participants, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Christina C Dieli-Conwright, PhD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Kang DW, Ficarra S, Wilson RL, Morgans AK, Nguyen PL, Rebbeck TR, Einstein DJ, Uno H, Mossanen M, Hill DM, Gonzalo-Encabo P, Norris MK, Gardiner J, Tjogas D, Greer J, Dieli-Conwright CM. Exercise to enhance cardiovascular health among black men with prostate cancer with androgen deprivation therapy (the POWER trial): A study protocol. Contemp Clin Trials. 2025 Aug;155:107973. doi: 10.1016/j.cct.2025.107973. Epub 2025 May 30. PMID 40451460